CLINICAL TRIAL: NCT03931785
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled, Parallel-group, Dose-range-finding Study of MD-7246 Administered Orally for 12 Weeks to Treat Abdominal Pain in Patients With Diarrhea-predominant Irritable Bowel Syndrome
Brief Title: A Study of MD-7246 to Treat Abdominal Pain in Patients With Diarrhea-predominant Irritable Bowel Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ironwood Pharmaceuticals, Inc. (Industry)
Collaborators: Allergan Sales, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MCP-103-205
Record Dates: First submitted 2019-04-22; First posted 2019-04-30 (Actual); Results first posted 2021-03-12 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-02

CONDITIONS: Irritable Bowel Syndrome With Diarrhea (IBS-D)
Keywords: Abdominal pain; Diarrhea; Irritable Bowel Syndrome
MeSH Terms: conditions — Abdominal Pain; Diarrhea; Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- MD-7246 300 μg (Experimental): 1 MD-7246 300-μg oral tablet and 3 matching placebo oral tablets
  Interventions: Drug: MD-7246; Drug: Placebo
- MD-7246 600 μg (Experimental): 2 MD-7246 300-μg oral tablets and 2 matching placebo oral tablets
  Interventions: Drug: MD-7246; Drug: Placebo
- MD-7246 1200 μg (Experimental): 4 MD-7246 300-μg oral tablets
  Interventions: Drug: MD-7246
- Placebo (Placebo Comparator): 4 matching placebo oral tablets
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MD-7246 — Oral tablet
  Arms: MD-7246 1200 μg; MD-7246 300 μg; MD-7246 600 μg
Drug: Placebo — Matching oral tablet
  Arms: MD-7246 300 μg; MD-7246 600 μg; Placebo

SUMMARY:
To evaluate the safety and tolerability, treatment effect on abdominal pain, and dose response of MD-7246 administered orally to patients with diarrhea-predominant irritable bowel syndrome (IBS-D).

ELIGIBILITY:
Inclusion Criteria:

* Patient meets the Rome IV criteria for diagnosis of IBS-D
* Patient maintains a minimum level of compliance with daily diary
* Female patients of childbearing potential must agree to use one of the following methods of birth control:

  1. Hormonal contraception
  2. Double-barrier method
  3. Maintenance of a monogamous relationship with a male partner who has been surgically sterilized by vasectomy

Exclusion Criteria:

* Patient has clinically significant findings on a physical examination and/or clinical laboratory tests
* Patient has symptoms of or been diagnosed with a medical condition that may contribute to abdominal pain
* Patient has a structural abnormality of the gastrointestinal (GI) tract or a disease or condition that can affect GI motility
* Patient has any protocol-excluded or clinically significant medical or surgical history that could confound the study assessments

NOTE: Additional inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 515 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wilmin Bartolini, PhD, Study Chair — Ironwood Pharmaceuticals, Inc.
Locations (79):
- United States (79):
  - Clinical Research Associates, Huntsville, Alabama
  - Elite Clinical Studies, Phoenix, Arizona
  - Arkansas Gastroenterology, North Little Rock, Arkansas
  - GW Research, Inc., Chula Vista, California
  - Kindred Medical Institute for Clinical Trials, LLC, Corona, California
  - Diagnamics Inc., Encinitas, California
  - St. Joseph Heritage Healthcare, Fullerton, California
  - Paragon Rx Clinical, Garden Grove, California
  - Grossmont Center For Clinical Research, La Mesa, California
  - Facey Medical Foundation, Mission Hills, California
  - Providence Clinical Research, North Hollywood, California
  - Precision Research Institute, San Diego, California
  - Paragon Rx Clinical, Inc. - Santa Ana, Santa Ana, California
  - UNISON Clinical Trials, Sherman Oaks, California
  - Millennium Clinical Trials, Thousand Oaks, California
  - Advanced Rx Clinical Research, Westminster, California
  - Peak Gastroenterology Associates, Colorado Springs, Colorado
  - Connecticut Clinical Research Institute, Bristol, Connecticut
  - Chase Medical Research of Greater New Haven LLC, Hamden, Connecticut
  - The Chappel Group Research, LLC, Kissimmee, Florida
  - Well Pharma Medical Research Corporation, Miami, Florida
  - New Horizon Research Center, Miami, Florida
  - San Marcus Research Clinic Inc, Miami Lakes, Florida
  - Ormond Medical Arts Pharmaceutical Research Center, Ormond Beach, Florida
  - Meridien Research, St. Petersburg, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Research Institute of Central Florida, LLC, Winter Park, Florida
  - Mount Vernon Clinical Research, LLC, Sandy Springs, Georgia
  - Rockford Gastroenterology Associates LTD, Rockford, Illinois
  - Clinical Trials Management LLC, Metairie, Louisiana
  - Clinical Trials of America -- LA LLC, West Monroe, Louisiana
  - Meritus Center For Clinical Research, Hagerstown, Maryland
  - Meridian Clinical Research, Rockville, Maryland
  - Boston Clinical Trials Inc, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - New England Center For Clinical Research Inc PrimaCare Research, LLC, Fall River, Massachusetts
  - MedVadis Research Corporation, Watertown, Massachusetts
  - Galen Research, Chesterfield, Missouri
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Barrett Clinic, P.C. - BTC - PPDS, La Vista, Nebraska
  - Meridian Clinical Research, Omaha, Nebraska
  - Clinical Research of South Nevada, Las Vegas, Nevada
  - Advanced Biomedical Research of America, Las Vegas, Nevada
  - Healthwise Medical Associates, Brooklyn, New York
  - Long Island Gastrointestinal Research Group LLP, Great Neck, New York
  - Rochester Clinical Research, Inc, Rochester, New York
  - Carolina Digestive Health Associates, Charlotte, North Carolina
  - Carolina Digestive Health Associates, Concord, North Carolina
  - Peters Medical Research, LLC, High Point, North Carolina
  - Clinical Trials of America-NC, LLC, Mount Airy, North Carolina
  - M3 Wake Research, Inc, Raleigh, North Carolina
  - PMG Research of Wilmington, Wilmington, North Carolina
  - Lyndhurst Clinical Research, Winston-Salem, North Carolina
  - PMG Research of Winston-Salem, Winston-Salem, North Carolina
  - Progressive Medicine of the Triad, LLC, Winston-Salem, North Carolina
  - Lillestol Research, Fargo, North Dakota
  - Hometown Urgent Care and Research, Cincinnati, Ohio
  - Hightop Medical Research Center, Cincinnati, Ohio
  - New Horizons Clinical Research, Cincinnati, Ohio
  - Hometown Urgent Care and Research, Columbus, Ohio
  - Remington Davis Inc, Columbus, Ohio
  - Hometown Urgent Care and Research, Dayton, Ohio
  - Central Sooner Research, Norman, Oklahoma
  - IPS Research Company, Oklahoma City, Oklahoma
  - Digestive Disease Specialists, Inc., Oklahoma City, Oklahoma
  - Oregon Center For Clinical Investigations Inc, Salem, Oregon
  - Partners In Clinical Research, Cumberland, Rhode Island
  - Ocean State Clinical Research Partners, Lincoln, Rhode Island
  - Mountain View Clinical Research Inc, Greer, South Carolina
  - WR-ClinSearch, LLC, Chattanooga, Tennessee
  - New Phase Research & Development, Knoxville, Tennessee
  - MW Clinical Research Center, Beaumont, Texas
  - Texas Tech University Health Sciences Center, El Paso, Texas
  - Southwest Clinical Trials, Houston, Texas
  - Quality Research Inc, San Antonio, Texas
  - Diagnostics Research Group, San Antonio, Texas
  - DCT - Stone Oak, LLC dba Discovery Clinical Trials, San Antonio, Texas
  - Advanced Research Institute, Ogden, Utah
  - New River Valley Research Institute, Christiansburg, Virginia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study included a Pretreatment Period, 14 to 21 days immediately before randomization. During this period, participants underwent symptomatic assessments in an electronic diary (eDiary); those who satisfied all entry criteria based on these assessments entered the Treatment Period and were randomized to 1 of 4 treatments: MD-7246 300, 600, or 1200 μg or placebo (1:1:1:1). Of the 515 participants in the Pretreatment Period, 127 were not randomized.
Groups:
- Placebo: 4 matching placebo oral tablets once daily (QD) for 12 weeks
- MD-7246 300 μg: 1 MD-7246 300-μg oral tablet and 3 matching placebo oral tablets QD for 12 weeks
- MD-7246 600 μg: 2 MD-7246 300-μg oral tablets and 2 matching placebo oral tablets QD for 12 weeks
- MD-7246 1200 μg: 4 MD-7246 300-μg oral tablets QD for 12 weeks
Period: Overall Study
Arm/Group | Placebo | MD-7246 300 μg | MD-7246 600 μg | MD-7246 1200 μg
Started | 97 | 97 | 97 | 97
Completed | 92 | 90 | 84 | 86
Not Completed | 5 | 7 | 13 | 11
Not completed — Lost to Follow-up | 4 | 1 | 4 | 3
Not completed — Adverse Event | 1 | 0 | 3 | 4
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Not completed — Noncompliance With Study drug | 0 | 1 | 0 | 0
Not completed — Other Not specified | 0 | 2 | 2 | 2
Not completed — Withdrawal by Subject | 0 | 2 | 4 | 1
Not completed — Pregnancy | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population: all participants who received at least one dose of study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | MD-7246 300 μg | MD-7246 600 μg | MD-7246 1200 μg | Total
Number analyzed (Participants) | 97 | 97 | 97 | 97 | 388
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.4 (13.12) | 45.0 (14.04) | 42.2 (14.38) | 45.1 (14.58) | 43.9 (14.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 63 | 67 | 68 | 264
  Male | 31 | 34 | 30 | 29 | 124
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 23 | 29 | 13 | 89
  Not Hispanic or Latino | 73 | 74 | 68 | 84 | 299
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 72 | 69 | 75 | 67 | 283
  Black or African American | 11 | 14 | 12 | 14 | 51
  Asian | 13 | 14 | 9 | 14 | 50
  Multiple Races | 0 | 0 | 1 | 2 | 3
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
Abdominal Pain at Its Worst at Each Week on a Numerical Rating Scale (NRS) [Mean (Standard Deviation); unit: units on a scale] — Abdominal pain is measured daily in an electronic diary (eDiary), using an 11-point NRS, where 0 is anchored with "no abdominal pain" and 10 is anchored with "worst possible abdominal pain." Baseline is derived from the eDiary data collected daily in the Pretreatment Period, specifically the period of time from 14 days before randomization up to the time of randomization.
  units on a scale | 6.22 (1.236) | 6.05 (1.112) | 5.95 (1.129) | 6.24 (1.169) | 6.12 (1.164)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Abdominal Pain at Its Worst on a NRS Through the Treatment Period
Description: Abdominal pain is measured daily in an eDiary, using an 11-point NRS, where 0 is anchored with "no abdominal pain" and 10 is anchored with "worst possible abdominal pain." The postbaseline weekly abdominal pain score is the average of the non-missing daily abdominal pain at its worst scores during a week (Weeks 1-12) if there are at least 4 daily scores entered into the eDiary during the week. Weekly change from baseline was calculated for each week as the weekly score minus the baseline score.
  Mixed model repeated measures (MMRM) results are based on a repeated measures analysis with treatment, analysis week, and treatment-by-week interaction as fixed effects and baseline as covariate. An unstructured covariance structure was used to model intra-subject correlation with subjects as a random effect.
  Baseline is derived from the eDiary data collected daily in the Pretreatment Period, specifically the period of time from 14 days before randomization up to the time of randomization.
Time Frame: Baseline, up to Week 12 (end of the Treatment Period)
Population: Modified Intent-to-Treat (mITT) Population: all randomized participants who received at least 1 dose of study drug. Participants with an assessment at Baseline and during the treatment period.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | MD-7246 300 μg | MD-7246 600 μg | MD-7246 1200 μg
Number analyzed (Participants) | 97 | 97 | 97 | 97
units on a scale | -2.01 (0.179) | -1.93 (0.179) | -1.58 (0.182) | -1.95 (0.180)
Statistical Analysis 1: Comparison: Placebo vs MD-7246 300 μg; Test type: Superiority; p = 0.7467, MMRM; Least squares (LS) mean difference = 0.08, 95% CI 2-sided [-0.42 to 0.58] — MD-7246 minus placebo
Statistical Analysis 2: Comparison: Placebo vs MD-7246 600 μg; Test type: Superiority; p = 0.0941, MMRM; LS mean difference = 0.43, 95% CI 2-sided [-0.07 to 0.93] — MD-7246 minus placebo
Statistical Analysis 3: Comparison: Placebo vs MD-7246 1200 μg; Test type: Superiority; p = 0.8098, MMRM; LS mean difference = 0.06, 95% CI 2-sided [-0.44 to 0.56] — MD-7246 minus placebo

2. Primary Outcome: Percentage of Participants Who Were 6/12 Week Abdominal Pain 30% Change Responders
Description: A 6/12 Week Abdominal Pain 30% Responder was a participant who had a decrease from baseline of ≥30% in the weekly abdominal pain score for that week for at least 6 out of the 12 weeks of the Treatment Period; for any week, a participant with < 4 daily abdominal pain scores available was considered a non-responder for that week.
  Abdominal pain is measured daily in an eDiary, using an 11-point NRS, where 0 is anchored with "no abdominal pain" and 10 is anchored with "worst possible abdominal pain." The postbaseline weekly abdominal pain score is the average of the non-missing daily abdominal pain at its worst scores during a week (Weeks 1-12) if there are at least 4 daily scores entered into the eDiary during the week.
Time Frame: Baseline through Week 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | MD-7246 300 μg | MD-7246 600 μg | MD-7246 1200 μg
Number analyzed (Participants) | 97 | 97 | 97 | 97
percentage of participants | 55.7 | 56.7 | 44.3 | 48.5
Statistical Analysis 1: Comparison: Placebo vs MD-7246 300 μg; Test type: Superiority; Difference in Responder Rate = 1.0, 95% CI 2-sided [-12.9 to 15.0] — Difference in responder rate (MD-7246 - placebo). 95% confidence intervals (CIs) for differences in responder rates were obtained using the normal approximation to the binomial distribution
Statistical Analysis 2: Comparison: Placebo vs MD-7246 600 μg; Test type: Superiority; Difference in Responder Rate = -11.3, 95% CI 2-sided [-25.3 to 2.6] — Difference in responder rate (MD-7246 - placebo). 95% CIs for differences in responder rates were obtained using the normal approximation to the binomial distribution
Statistical Analysis 3: Comparison: Placebo vs MD-7246 1200 μg; Test type: Superiority; Difference in Responder Rate = -7.2, 95% CI 2-sided [-21.2 to 6.8] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 4: Comparison: Placebo vs MD-7246 300 μg; Test type: Superiority; p = 0.8852, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.043, 95% CI 2-sided [0.591 to 1.839] — Odds ratio for response (MD-7246 : placebo)
Statistical Analysis 5: Comparison: Placebo vs MD-7246 600 μg; Test type: Superiority; p = 0.1152, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.634, 95% CI 2-sided [0.360 to 1.117] — Odds ratio for response (MD-7246 : placebo)
Statistical Analysis 6: Comparison: Placebo vs MD-7246 1200 μg; Test type: Superiority; p = 0.3157, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.749, 95% CI 2-sided [0.425 to 1.317] — Odds ratio for response (MD-7246 : placebo)

ADVERSE EVENTS:
Time Frame: From the first dose of double-blind study drug and within 1 day of the date of last dose of double-blind study drug in the treatment period (up to Week 12 / Day 85). Mean treatment duration was 82.8, 77.3, and 80.8 days in the MD-7246 300, 600, and 1200 μg groups, respectively, and 83.3 days in the placebo group.
Arm/Group | Placebo | MD-7246 300 μg | MD-7246 600 μg | MD-7246 1200 μg
All-Cause Mortality (participants affected / at risk) | 0/97 | 0/97 | 0/97 | 0/97
Serious Adverse Events (participants affected / at risk) | 0/97 | 0/97 | 0/97 | 1/97
Other Adverse Events (participants affected / at risk) | 27/97 | 28/97 | 42/97 | 52/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=97) | MD-7246 300 μg (N=97) | MD-7246 600 μg (N=97) | MD-7246 1200 μg (N=97)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | NA | NA | NA | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=97) | MD-7246 300 μg (N=97) | MD-7246 600 μg (N=97) | MD-7246 1200 μg (N=97)
Nasopharyngitis (Infections and infestations) | 4 | 5 | 5 | 3
Headache (Nervous system disorders) | 2 | 4 | 4 | 4
Nausea (Gastrointestinal disorders) | 1 | 3 | 3 | 4
Upper respiratory tract infection (Infections and infestations) | 7 | 1 | 3 | 5
Influenza (Infections and infestations) | 1 | 1 | 1 | 5
Constipation (Gastrointestinal disorders) | 2 | 1 | 3 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 4 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 2 | 2
Sinusitis (Infections and infestations) | 1 | 1 | 0 | 4
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 1
Urinary tract infection (Infections and infestations) | 3 | 1 | 2 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0 | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 2 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 2
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 2 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 2 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 0
Hypertension (Vascular disorders) | 1 | 2 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 2 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Bacterial vaginosis (Infections and infestations) | 0 | 0 | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI may publish or disclose the results of the study 24 months after final data lock provided that sponsor can review the publication prior to public release, sponsor can request removal of confidential information of sponsor (not including results of trial), and sponsor can request a publication delay in order to protect potentially patentable information. Furthermore, if a publication committee is developing an initial publication, PI is to delay disclosure until that publication is published.

DOCUMENTS (2):
  • Study Protocol (2019-01-29): https://cdn.clinicaltrials.gov/large-docs/85/NCT03931785/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-14): https://cdn.clinicaltrials.gov/large-docs/85/NCT03931785/SAP_001.pdf